CLINICAL TRIAL: NCT05171309
Title: Camrelizumab in Combination With Apatinib Plus NK Cell in Patients With Advanced Hepatocellular Carcinoma (CAN): A First-line, Phase-II, Single-arm Trial
Brief Title: Camrelizumab in Combination With Apatinib Plus NK Cell for Advanced HCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2021-372
Record Dates: First submitted 2021-12-26; First posted 2021-12-28 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Camrelizumab; Apatinib; NK cell
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — apatinib; camrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab in combination with apatinib plus NK cell (Experimental): Drug: Apatinib 250 mg once daily (QD) oral dosing.
  Other Names:
  • Apatinib Drug: Camrelizumab 200 mg intravenously every 2 weeks.
  Other Names:
  • Camrelizumab Drug: NK cell Cord blood derived NK cells 4 cycles, one cycle is defined as: total cells ≥1×109 per time, continuous intravenous infusion for 2 days every 14±2 days
  Interventions: Drug: Apatinib; Drug: Camrelizumab; Drug: NK cell

INTERVENTIONS:
Drug: Apatinib — 250 mg once daily (QD) oral dosing.
Drug: Camrelizumab — 200 mg intravenously every 2 weeks.
Drug: NK cell — Cord blood derived NK cells 4 cycles, one cycle is defined as: total cells ≥1×109 per time, continuous intravenous infusion for 2 days every 14±2 days

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Camrelizumab in combination with apatinib plus NK cell in patients with advanced hepatocellular carcinoma.

DETAILED DESCRIPTION:
The IMbrave150 study has demonstrated a new regimen to be superior to sorafenib by reducing 42% of death risk, making "T+A" strategy to be the first-line treatment for patients with advanced HCC. Meanwhile, the RESCUE research showed that combined camrelizumab with apatinib has promising objective response rate (ORR=34.3%) and disease control rate (DCR=77.1%) in advanced HCC patients as first-line treatment. Nevertheless, the above researches both show only a fraction of patients benefits from the anti-PD-1/PD-L1 in combination with antiangiogenic therapy. Therefore, it's urgently needed to explore better combinational strategies with other treatments to enhance the efficacy of anti-PD-1 in combination with antiangiogenic therapy. Recently, Pembrolizumab plus allogeneic NK cells have been proved to be effective in advanced non-small cell lung cancer patients. However, there is no study available now analyzing the efficacy and safety of Camrelizumab in combination with apatinib plus NK cell in patients with advanced hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 ≤ 70, male or female;
2. Clinical or pathologically confirmed BCLC B (tumor numbers ≥ 4) or C stage hepatocellular carcinoma (except intracranial metastasis);
3. At least one intrahepatic evaluable tumor existed, intrahepatic tumor is the primary tumor burden (according to RECIST v1.1, the long diameter of spiral CT scan of the measurable lesion is ≥ 10 mm or the short diameter of enlarged lymph nodes is ≥ 15 mm);
4. No previous systematic (including systematic study drugs) HCC treatment;
5. No contraindications of carrizumab, apatinib and NK cell therapy;
6. Patients who have previously received local treatment (such as microwave ablation, radiofrequency ablation, absolute ethanol or acetic acid injection, cryoablation, high intensity focused ultrasound, transcatheter arterial chemoembolization or perfusion chemotherapy, etc.), A. if the focus has not received local treatment before, it can be used as the target focus; b. If the focus has received local treatment before, it can be used as the target focus after the progress is evaluated according to RECIST v1.1 standard;
7. Child-Pugh score small or equal to 7 points (Child-Pugh A-B);
8. Life expectancy of at least 12 weeks;
9. ECOG score: 0 to 1 (according to the ECOG score classification);
10. The subjects voluntarily joined the study, signed the informed consent form, had good compliance and cooperated with the follow-up;
11. For female that non-surgical sterilization or in childbearing age need to use a medically approved contraceptive (such as an intrauterine device, contraceptive or condom) during the study period and within 3 months after the end of the study treatment period; For female that non-surgical sterilization or in childbearing age must have a negative serum or urine HCG test within 72 hours prior to study enrollment; and must be nonlactating; for male patients whose partner in a childbearing age, effective methods of contraception should be given during the trial and at the end of Camrelizumab injection.
12. The laboratory parameters meets the following requirements (no blood components and cell growth factors are allowed within 14 days before the first dose):

    Absolute neutrophil count ≥ 1.5 × 109 / L; Platelets ≥ 50 × 109 / L; Hemoglobin ≥ 80 g / L; Biochemical examination shall meet the following standards: TBIL < 1.5 × ULN； ALT and AST < 5 × ULN； Bun and Cr ≤ 1 × The clearance rate of ULN or endogenous creatinine ≥ 50ml / min (Cockcroft Gault formula).

    Stable coagulation function: INR ≤ 1.5, PTT < 1.2 times the upper limit of normal value (except for tumor related anticoagulant therapy).
13. Anti HBV therapy should be initiated before enrollment for patients with detectable HBV DNA.

Exclusion Criteria:

1. Accepted any systematic treatment before (excluding traditional Chinese medicine and traditional Chinese medicine preparations);
2. Existed Hepatobiliary carcinoma, sarcomatoid HCC, mixed cell carcinoma and fibrous lamellar cell carcinoma; Active malignant tumors other than HCC within 5 years or at the same time. Limited localized tumors, such as basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, prostate cancer in situ, in situ carcinoma of the cervix, and breast cancer in situ, can be included.
3. History of organ allograft;
4. Moderate and severe ascites with clinical symptoms, i.e. those who need therapeutic puncture and drainage, or child Pugh score > 2 (except those who only show a small amount of ascites on imaging but are not accompanied by clinical symptoms); Uncontrolled or moderate pleural effusion and pericardial effusion;
5. With a history of gastrointestinal bleeding or definite tendency of gastrointestinal bleeding within 6 months before enrollment, such as bleeding risk or severe esophageal and gastric varices, local active gastrointestinal ulcer lesions, and positive continuous fecal occult blood, shall not be included in the group (if fecal occult blood is positive in the baseline period, it can be rechecked. If it is still positive after recheck, gastroduodenoscopy is required (EGD), if EGD indicates the risk of bleeding, esophageal and gastric varices cannot be included in the group);
6. Abdominal fistula, gastrointestinal perforation or abdominal abscess occurred within 6 months before the start of the study drug;
7. Events of arterial/venous thrombosis occurring within the first 6 months of enrollment, such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism;
8. Aspirin (> 325 mg / day (maximum antiplatelet dose) or dipyridamole, ticlopidine, clopidogrel and cilostazol were currently or recently used (within 10 days before the start of study treatment);
9. hrombosis or embolism events occurred within 6 months before the start of the study drug, such as cerebrovascular accidents (including transient ischemic attack, intracerebral hemorrhage, cerebral infarction), pulmonary embolism, etc;
10. Suffering heart diseases with clinical symptoms or those not well controlled, such as: (1) heart failure in NYHA class 2 or higher; (2) unstable angina; (3) myocardial infarction occurred within 1 year; (4) clinically symptomatic supraventricular or ventricular arrhythmia requiring treatment or intervention; (5) Tc > 450ms (male); QTc > 470ms (female);
11. Suffering from hypertension, and cannot be well controlled by antihypertensive drugs (systolic blood pressure ≥ 140mmHg or diastolic blood pressure ≥90 mmHg);
12. Major vascular diseases (e.g., aortic aneurysms requiring surgical repair or recent peripheral arterial thrombosis) occurred within 6 months before the start of the study drug;
13. Severe, unhealed or cracked wounds and active ulcers or untreated fractures;
14. Major surgical treatment (except diagnosis) within 4 weeks before the start of study treatment or major surgical treatment is expected during the study period;
15. Inability to swallow tablets, malabsorption syndrome, or any condition affecting gastrointestinal absorption;
16. Clinical signs or symptoms of intestinal obstruction and / or gastrointestinal obstruction within 6 months before the start of study treatment, including incomplete obstruction related to original disease or requiring routine parenteral hydration, parenteral nutrition or tube feeding:
17. At the initial diagnosis, patients with incomplete obstruction / obstruction syndrome / signs / symptoms of intestinal obstruction may be admitted to the study if they receive definite (surgical) treatment to subside the symptoms;
18. There is evidence of intraabdominal pneumatosis that cannot be explained by puncture or recent surgery;
19. Known central nervous system tumors including metastatic brain disease;
20. Metastatic diseases involving major airways or blood vessels (such as portal vein trunk or vena cava completely occluded due to tumor invasion, which refers to the confluence of splenic vein and superior mesenteric vein and the branches of hepatic portal vein divided into left and right branches) or large mediastinal tumor mass in the center (less than 30 mm from the ridge);
21. With a history of hepatic encephalopathy;
22. Present with interstitial pneumonia or interstitial lung disease, or previous history of interstitial pneumonia or interstitial lung disease requiring hormone treatment, or other pulmonary fibrosis, organic pneumonia (e.g., bronchiolitis obliterans), pneumoconiosis, drug-related pneumonia, idiopathic pneumonia or chest computed tomography in the screening period that may interfere with the judgment and treatment of immune-related pulmonary toxicity (CT) subjects with evidence of active pneumonia or severely impaired pulmonary function on the figure, allowed radiation field to have radiation pneumonia; active tuberculosis;
23. The patient has any active auto-immune disease or a history of autoimmune disease;
24. immunosuppressive treatment with immunosuppressants or systemic hormones within 14 days before the start of study treatment (dose > 10mg / day prednisone or other equivalent hormones);
25. Applying strong CYP3A4 / CYP2C19 inducers including rifampicin (and its analogues) and Hypericum perforatum or strong CYP3A4 / CYP2C19 inhibitors within 14 days before the start of study treatment;
26. Severe infection within 4 weeks before the start of study treatment, including but not limited to hospitalization due to complications of infection, bacteremia or severe pneumonia; oral or intravenous administration of therapeutic antibiotics within 2 weeks before the start of study treatment (patients receiving prophylactic antibiotics (e.g. prevention of urinary tract infection or exacerbation of chronic obstructive pulmonary disease are eligible to participate in the study);
27. Known history of HIV;
28. Co-infection of hepatitis B and HCV.
29. Patients have previously received other anti-PD-1 antibody therapy or other immunotherapy against PD-1/PD-L1, or have received apatinib before;
30. Palliative radiotherapy for non target lesions allowed to control symptoms must be completed at least 2 weeks before the start of study treatment, and the adverse events caused by radiotherapy have not recovered to ≤ CTCAE level 1.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | From date of first dose of study drug until disease progression, development of unacceptable toxicity, withdrawal of consent, or sponsor termination (up to approximately 3 years)
  ORR is defined as the percentage of participants who have best overall response (BOR) of complete response (CR) or partial response (PR) at the time of data cutoff as assessed by RECIST 1.1

SECONDARY OUTCOMES:
The disease control rate (DCR) | From date of first dose of study drug until disease progression, stable disease, development of unacceptable toxicity, withdrawal of consent, or sponsor termination (up to approximately 3 years)
  DCR is defined as the percentage of participants who have best overall response (BOR) of complete response (CR) or partial response (PR) or stable disease (SD) at the time of data cutoff as assessed by RECIST 1.1
The median progression free survival time (mPFS) | From date of first dose of study drug to the date of first documentation of disease progression (up to approximately 3 years)
  The progression free survival time (mPFS) defined as the time from the first study dose date to the date of first documentation of disease progression as assessed by RECIST 1.1
The median overall survival time (mOS) | From the start date of the Treatment Phase until date of death from any cause (up to approximately 3 years)
  OS is measured from the start date of the Treatment Phase (date of first study dose) until date of death from any cause. Participants who are lost to follow-up and the participants who are alive at the date of data cutoff will be censored at the date the participant was last known alive or the cut-off date, whichever comes earlier.
Progression free survival rate at 12 months | From date of first dose of study drug to the date of first documentation of disease progression or death, whichever occurs first (up to approximately 3 years)
  The progression free survival time defined as the time from the first study dose date to the date of first documentation of disease progression as assessed by RECIST 1.1
Overall survival rate at 12 months | From date of first dose of study drug to the date of first documentation of death from any cause, whichever occurs first (up to approximately 3 years)
  OS is measured from the start date of the Treatment Phase (date of first study dose) until date of death from any cause. Participants who are lost to follow-up and the participants who are alive at the date of data cutoff will be censored at the date the participant was last known alive or the cut-off date, whichever comes earlier.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | From the start date of the Treatment Phase until date of death from any cause (up to approximately 3 years)
  Safety will be evaluated according to the NCI CTCAE Version 5.0. All observations pertinent to the safety of the study medication will be recorded on the CRF and included in the final report.

CONTACTS AND LOCATIONS:
Overall Officials: Jinzhang Chen, MD., Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No